CLINICAL TRIAL: NCT04689282
Title: Safety/Efficacy of Intranasally-Administered Bioactive Factors Produced by M2 Type Macrophages in Children With Developmental Speech Disorders
Brief Title: Intranasal Inhalations of M2 Macrophage Soluble Factors in Children With Developmental Speech Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alexander A Ostanin, Head of Clinical Department, Russian Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCI-23/06/2017
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Language Delay; Language; Developmental Disorder, Expressive; Language; Developmental Disorder, Receptive; Autism Spectrum Disorder; Attention Deficit-Hyperactivity Disorder; Speech Disorders in Children
Keywords: M2 type macrophages; Cytokines; Intranasal administration; Neuroprotection; neuroregeneration; Speech disorders
MeSH Terms: conditions — Language Development Disorders; Language; Developmental Disabilities; Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Speech Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intranasal M2-BFs (Experimental): Intranasally-Administered Bioactive Factors, Produced by M2 Type Macrophages (M2-BFs). M2 were generated in vitro from peripheral blood of a parent during 7 days. Cell-free culture medium, containing M2-BFs, was collected, and aliquots of 2 mL/vial were cryopreserved.
  30 children with speech disorders will receive their first doses (n=2-3) of M2-BFs in Clinic and wait 2 hrs to determine any short-time adverse effects of inhaled dose. The subsequent course of intranasal inhalations (once a day up to 30 days) performed as outpatient treatment.
  Interventions: Biological: Bioactive Factors, Produced by M2 Type Macrophages (M2-BFs).

INTERVENTIONS:
Biological: Bioactive Factors, Produced by M2 Type Macrophages (M2-BFs). — Intranasal delivery of M2-BFs is performed with the aerosol inhaler device (nebulizer), 2.0 mL once a day up to 30 days.

SUMMARY:
The investigators have designed an innovative proof-of-concept trial designed to provide data as to whether the speech difficulties in children with developmental dysphasia (DD) are improved with intranasal inhalations of bioactive factors (BF), produced by macrophages of M2 phenotype (M2-BFs). The rationale for this approach is the ability of central nervous system (CNS) to repair and the important role of macrophages in the regulation of this process. It was found that type 2 macrophages (M2) have anti-inflammatory and neurorestorative potential, in contrast to pro-inflammatory and neurotoxic effects of М1 cells. The influence of M2 is largely realized through the production of a wide spectrum of bioactive factors (cytokines, chemokines, growth factors, neuropeptides, microvesicles etc) that inhibit inflammation, protect neurons from apoptosis, stimulate neurogenesis, the growth and remyelination of axons, the formation of new synapses and activate angiogenesis. This study uses M2-BFs, as therapeutic tool, and intranasal administration focusing on nose to brain transport, as a mode of delivery. Expected clinical effects in treated children: improvement of speech understanding, word formation, grammatical structure of speech and formation of coherent speech.

DETAILED DESCRIPTION:
Neuroinflammation plays a central role in the pathogenesis of any damage to the central nervous system (CNS) profoundly affecting the ability of neural cells to survive and to regenerate. Macrophages play a key role in the regulation of neuroinflammation, but their role is ambiguous. In fact, macrophages can both induce neuronal and glial toxicity and promote tissue repair. The opposite effects of macrophages are largely due to their plasticity and functional heterogeneity. Thus, classical pro-inflammatory macrophages (M1) are tissue-destructive, while anti-inflammatory (M2) macrophages mediate tissue repair. In addition, M2 predominantly induce the Th2 response, which is particularly beneficial in CNS repair. Using low serum conditions the investigators have generated M2-like macrophages and evaluated their phenotypic and functional features [1]. The data indicate that M2, in contrast to pro-inflammatory M1, produced significantly lower levels of pro-inflammatory cytokines (IL-1β, tumor necrosis factor-α, IL-6, IL-18, IL-12), chemokines (IL-8, monocyte chemoattractant protein 1-1) and Th1/Th2-cytokines (interferon-γ, IL-2, IL-4) coupled with a high IL-10 level. M2 were capable of producing neurotrophic (brain-derived neurotrophic factor, insulin-like growth factor-1), angiogenic (vascular endothelial growth factor), and other growth factors (erythropoietin, granulocyte-colony stimulating factor, basic fibroblast growth factor, epidermal growth factor) with neuroprotective and regenerative activity.

Pilot clinical trials have demonstrated the safety and clinical efficacy of intrathecal administration of M2 in children with severe cerebral palsy [2, 3] and in nonacute stroke patients [4]. Moreover, intranasal delivery of M2 macrophage-derived soluble products reduces neuropsychological deficit in patients with cerebrovascular disease [5]. Given this data, the investigators expect that intranasal administration of the M2-BFs (Bioactive Factors) will reduce the severity of speech disorders in children, including improving speech understanding, sensorimotor speech level, word formation skills, as well as the formation of the grammatical structure of speech and coherent speech. Of note, intranasal administration of M2 soluble factors allow to delivery bioactive agents to brain through the olfactory and trigeminal ways across brain-blood barrier.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-18
* Speech disorders verified by speech therapist and neurologist
* Adequate hearing/vision to follow conversation
* Russian speaker
* A written informed consent of the parents/close relatives

Exclusion Criteria:

* Acute infectious disease (bacterial, fungal, or viral)
* Seizures
* Intolerance to gentamicin and/or multiple drug allergies
* Participation in other clinical trials

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in the severity of speech disorders according to Speech Assessment Scale (SAS) | Baseline and 6 months after treatment
  Speech Assessment Scale (SAS) is used to assess language development in children in six functional domains: Speech Comprehension; Sensomotor speech level; Grammatical structure of speech and inflection; Vocabulary and vocabulary skills; Connected speech; Gross and fine motor skills. Max total score:160 points (units of scale). Clinical improvement is manifested in an enhancement in the SAS score.

SECONDARY OUTCOMES:
The number of patients with adverse events | up to 6 months after treatment
  Occurrence of adverse events including allergic, toxic, inflammatory reactions; neurological worsening; seizures

CONTACTS AND LOCATIONS:
Overall Officials: Elena R Chernykh, MD, PhD, Study Chair — Institute of Fundamental and Clinical Immunology; Alexander A Ostanin, MD, PhD, Principal Investigator — Institute of Fundamental and Clinical Immunology
Locations (1):
- Institute of Fundamental and Clinical Immunology, Novosibirsk, Russia

REFERENCES:
- [Background] Sakhno LV, Shevela EY, Tikhonova MA, Ostanin AA, Chernykh ER. The Phenotypic and Functional Features of Human M2 Macrophages Generated Under Low Serum Conditions. Scand J Immunol. 2016 Feb;83(2):151-9. doi: 10.1111/sji.12401. PMID 26678544
- [Background] Chernykh ER, Kafanova MY, Shevela EY, Sirota SI, Adonina EI, Sakhno LV, Ostanin AA, Kozlov VV. Clinical experience with autologous M2 macrophages in children with severe cerebral palsy. Cell Transplant. 2014;23 Suppl 1:S97-104. doi: 10.3727/096368914X684925. Epub 2014 Oct 9. PMID 25302537
- [Background] Chernykh ER, Shevela EYa, Kafanova MYu, Sakhno LV, Polovnikov EV, Ostanin AA. Monocyte-derived macrophages for treatment of cerebral palsy: a study of 57 cases. J Neurorestoratology. 2018; 6: 41-47. doi.org/10.2147/JN.S158843
- [Background] Chernykh ER, Shevela EY, Starostina NM, Morozov SA, Davydova MN, Menyaeva EV, Ostanin AA. Safety and Therapeutic Potential of M2 Macrophages in Stroke Treatment. Cell Transplant. 2016;25(8):1461-71. doi: 10.3727/096368915X690279. Epub 2015 Dec 14. PMID 26671426
- [Background] Shevela E, Davydova M, Starostina N, Yankovskaya A, Ostanin A, Chernykh E. Intranasal delivery of M2 macrophage-derived soluble products reduces neuropsychological deficit in patients with cerebrovascular disease: a pilot study. J Neurorestoratology. 2019; 7: 89-100. doi:10.26599/JNR.2019.9040010
- See also: Shevela E.Y., et al. Therapeutic effect of soluble factors of M2 phenotype macrophages in children with language impairments. Medical Immunology (Russia). 2021;23(5):1137-1150. (In Russ.) https://doi.org/10.15789/1563-0625-TEO-2224 — https://doi.org/10.15789/1563-0625-TEO-2224